CLINICAL TRIAL: NCT05372874
Title: Evaluation of the Effect of Direct-Acting Antiviral Agents on Melatonin Level in Chronic Hepatitis C Patients in Egypt.
Brief Title: Treatment of Hepatitis c by Using Direct-acting Antiviral
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Heba Mohammed Hashem Ali, Assistant lecturer, Tanta University
Other Study IDs: Hepatitis C
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy voluntaries control group (Group 1)
- sofosbuvir/daclatasvir treated group (group 2)
  Interventions: Drug: Direct Acting Antivirals
- sofosbuvir /daclatasvir/ ribavirin treated group (group 3)
  Interventions: Drug: Direct Acting Antivirals

INTERVENTIONS:
Drug: Direct Acting Antivirals — hepatitis C patients will be treated by direct acting antiviral drugs (DAAs)for 12 weeks.
  Groups: sofosbuvir /daclatasvir/ ribavirin treated group (group 3); sofosbuvir/daclatasvir treated group (group 2)

SUMMARY:
Patients with hepatitis c showed increased level of oxidative stress. Increased level of serum lipid peroxidation leads to the production of toxic mediators as malondialdehyde (MDA) which lead to disease progression. Chronic stress shunt tryptophan which is essential amino acid toward kynurenic pathway leading to lower level of serotonin and melatonin level. Currently, direct-acting antivirals (DAAs) show well-established efficacy against hepatitis C virus (HCV).

ELIGIBILITY:
Inclusion Criteria:

* chronic hepatitis C patients had no other cause of liver disease

Exclusion Criteria:

* Patients with hepatitis B virus (HBV).
* Patients with acute hepatitis.
* Patients with renal insufficiency.
* Patients with Hepatocellular carcinoma (HCC) or other types of malignancy.
* Patients on current use of melatonin.
* Patients using of any of medications that have interaction with melatonin.
* Patients work in night shifts.
* Patients are consuming a lot of caffeine or heavy smokers.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatitis C patients treated by daclatasvir/sofosbuvir or sofosbuvir /daclatasvir/ ribavirin.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-05-06 (Estimated); Primary Completion 2022-07-12 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in malondialdehyde (MDA) level. | 12 weeks following end of treatment.
  Malondialdehyde (MDA) levels will be measured by the TBARS assay (thiobarbituric acid reactive substance assay)
Change in melatonin level. | 12 weeks following end of treatment.
  Melatonin will be measured by using immunological method.

CONTACTS AND LOCATIONS:
Overall Officials: Sabry A AbouSaif, Professor, Principal Investigator — Tanta University; Sally E Abu-Risha, Associate professor, Principal Investigator — Tanta University; Medhat I Abd-El Hamed, Professor, Principal Investigator — Faculty of Medicine, Al-Azhar University

IPD SHARING:
Plan to Share IPD: Undecided